CLINICAL TRIAL: NCT02132624
Title: CD19-targeting 3rd Generation CAR T Cells for Refractory B Cell Malignancy - a Phase I/IIa Trial.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Karolinska University Hospital (Other); AFA Insurance (Industry); Swedish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003:TCELL; 2013-001393-19 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: B Cell Lymphoma; B Cell Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR T cells (Experimental): Autologous 3rd generation CD19-targeting CAR T cells
  Interventions: Biological: Autologous 3rd generation CD19-targeting CAR T cells

INTERVENTIONS:
Biological: Autologous 3rd generation CD19-targeting CAR T cells — Autologous CD19-targeting CAR T cells with three signaling domains derived from CD3zeta, CD28 and 4-1BB.

SUMMARY:
Chimeric antigen receptor (CAR) T cells targeting CD19 will be evaluated for safety and efficacy in patients with B cell lymphoma or leukemia. The CAR consists of a CD19 targeting antibody scFv with three intracellular signaling domains derived from CD3 zeta, CD28 and 4-1BB. Autologous T cells will be gene engineered with the CAR gene using a retrovirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD19+ B-cell lymphoma or leukemia.
* Measurable disease.
* Performance status ECOG 0-2.
* >18 years old.
* Fertile females/males must consent to use contraceptives during participation of the trial.
* Signed informed consent.

Exclusion Criteria:

* Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
* Patients with primary CNS lymphoma.
* Known human immunodeficiency virus (HIV) infection.
* Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection).
* Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient.
* Treatment with an investigational product within 30 days prior to enrollment, or at least 5 half lives of that drug, which is longest.
* Patients that do not consent to that tissue and blood samples are stored in a biobank.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
CAR T cell persistence | At week 1 and 5, there after every 3 months post treatment up to 24 months
  Presence of circulating CAR T cells will be evaluated with flow cytometry and real time PCR in patient blood.

SECONDARY OUTCOMES:
Tumor load | Every 3 months post treatment up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

OTHER OUTCOMES:
B cell number and immunoglobulins | Weekly for 5 weeks, then every 3 months post treatment up to 24 months
  Number of blood B cells and immunoglobulins will be evaluated by routine diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Loskog, PhD, Study Director — Uppsala University; Gunilla Enblad, MD, PhD, Principal Investigator — Uppsala University Hospital; Hans Hagberg, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Dept of Oncology, Uppsala, Sweden

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Enblad G, Karlsson H, Gammelgard G, Wenthe J, Lovgren T, Amini RM, Wikstrom KI, Essand M, Savoldo B, Hallbook H, Hoglund M, Dotti G, Brenner MK, Hagberg H, Loskog A. A Phase I/IIa Trial Using CD19-Targeted Third-Generation CAR T Cells for Lymphoma and Leukemia. Clin Cancer Res. 2018 Dec 15;24(24):6185-6194. doi: 10.1158/1078-0432.CCR-18-0426. Epub 2018 Aug 10. PMID 30097433